CLINICAL TRIAL: NCT03592576
Title: Expanded Access to Navitoclax
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C19-199; C19-922 (Other: AbbVie)
Record Dates: First submitted 2018-07-10; First posted 2018-07-19 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Myelofibrosis; Acute Lymphocytic Leukemia (ALL); Lymphoblastic Lymphoma
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — navitoclax; venetoclax

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Navitoclax — Tablet, Oral
  Other Names: ABT-263
Drug: Venetoclax — Tablet, Oral
  Other Names: Venclexta; ABT-199; GDC-0199

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to navitoclax prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

Min Age: 4 Years | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult